CLINICAL TRIAL: NCT05269914
Title: Safety, Efficacy and Pharmacokinetics of XKDCT023 in Adult Patients With Recurrent or Refractory Diffuse Large B-cell Lymphoma
Brief Title: Safety, Efficacy and Pharmacokinetics of XKDCT023 in DLBCL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XKDCT023-DLBCL
Record Dates: First submitted 2021-12-03; First posted 2022-03-08 (Actual); Last update posted 2022-03-08 (Actual); Status verified 2022-03

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse large B-cell lymphoma; Autologous anti-CD19 CAR-T cells
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Intervention Model Description: Single infusion of autologous anti-CD19 car-t cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous anti-CD19 CAR-T cell injection (Experimental): with 1.00×106 CAR+T cells/kg, 3.00×106 CAR+T cells /kg and 9.00×106 CAR+T cells/kg
  Interventions: Other: Autologous anti-CD19 CAR-T cell injection

INTERVENTIONS:
Other: Autologous anti-CD19 CAR-T cell injection — According to preclinical research, existing preliminary clinical data and similar approved therapeutic products (kte-c19 of Kate company, the trade name is yescarta ®） According to the clinical trial results, three doses (the number of cells per unit body weight) were selected as the therapeutic dose of this study. Among the patients who increased the dose according to the "3 + 3" design, the number of target cells in each dose group was: (1) the first dose group was 1.00 × 106 Car + T cells / kg, 20% dose error is allowed. (2) the second dose group is 3.00 × 106 Car + T cells / kg, 20% dose error is allowed. (3) the third dose group is 9.00 × 106 Car + T cells / kg, 20% dose error is allowed.

SUMMARY:
This study is a phase I multicenter, single arm, open, dose increasing, single treatment clinical study. This study plans to recruit a total of about 10-16 adult patients with CD19 positive recurrent or refractory DLBCL for a single autologous car-t cell therapy. There are three dose groups in the study. The first dose group has one patient. If there is no dose limiting toxicity (DLT), it can be increased to the second dose group, otherwise it will continue to be enrolled according to the "3 + 3" method; The follow-up dose group is conducted according to the traditional "3 + 3" design, that is, three subjects are first enrolled in a dose group. If there is no dose limiting toxicity (DLT) in the three patients in the dose group, it can be increased to the next higher dose after completing the DLT observation period; If DLT occurs in 1 of the 3 patients in the dose group, it is necessary to continue to enroll 3 patients in the dose group for DLT observation. The highest dose level of DLT in less than or equal to 1 of the last 6 confirmed patients will be defined as MTD. The safety of car-t treatment was evaluated by observing the adverse events after cell therapy; Evaluate the effectiveness of car-t treatment compared with the results or historical data of the patient's own previous standard treatment regimen. Blood and bone marrow were collected before and 12 months after cell infusion, the number and activity of car-t cells were detected, and the pharmacokinetics (PK) of car-t cells was evaluated.

DETAILED DESCRIPTION:
This study is a phase I multicenter, single arm, open, dose increasing, single treatment clinical study. This study plans to recruit a total of about 10-16 adult patients with CD19 positive recurrent or refractory DLBCL for a single autologous car-t cell therapy. There were three dose groups in the study, and one patient in the first dose group, If there is no dose limiting toxicity (DLT), it can be increased to the second dose group, otherwise it will continue to be included in the group according to the "3 + 3" method; the follow-up dose group is designed according to the traditional "3 + 3" design, that is, three subjects will be included in a dose group first, if there is no dose limiting toxicity in the three patients in the dose group (DLT), after completing the DLT observation period, it can be increased to the next higher dose; if one of the three patients in the dose group has DLT, it is necessary to continue to join the group of three patients in the dose group for DLT observation. The highest dose level of DLT in less than or equal to one of the six patients finally confirmed will be defined as MTD. By observing the adverse events after cell therapy, the patients will be evaluated Evaluate the safety of car-t treatment; Evaluate the effectiveness of car-t treatment compared with the results or historical data of the patient's own previous standard treatment regimen. Blood and bone marrow were collected before and 12 months after cell infusion to detect the number and activity of car-t cells, Evaluate the pharmacokinetics (PK) of car-t cells. During the study, the blood samples used for the production of car-t cells will be transported to Shenzhen xiankangda Life Sciences Co., Ltd. (sponsor). After the production of car-t cells is completed, the car-t cells will be sent to the research unit so that the researchers can infuse them to the corresponding subjects.

ELIGIBILITY:
Inclusion Criteria:

* All subjects or legal guardians must sign the informed consent approved by the ethics committee in writing before starting any screening procedure.
* Adult patients aged 18 and over with recurrent or refractory DLBCL.
* Bone marrow negative or bone marrow lymphoma cells in screening stage determined by CT scan < 30%.
* The subject had been adequately treated before.
* According to the revised IWG malignant lymphatic efficacy evaluation criteria (2007 Edition), there was at least one measurable lesion in the baseline period.
* Estimated survival ≥ 12 weeks.
* The baseline ECoG score was 0 or 1.
* Adequate organ function.
* Hemodynamics determined by echocardiography or multichannel radionuclide angiography (MUGA) were stable and left ventricular ejection fraction (LVEF) ≥ 45%.
* Sufficient bone marrow reserve without blood transfusion.
* There must be non mobilized apheresis or peripheral blood collected cells for car-t cell production.
* According to the judgment of the researcher, the patient has fully recovered from the toxicity of previous anti-tumor treatment and is suitable for pretreatment chemotherapy and car-t cell treatment.
* Women of childbearing age and all male subjects must agree to use efficient contraceptive methods until at least 12 months after xkdct023 infusion, and until two consecutive PCR tests show that car-t cells are no longer present in the body.

Exclusion Criteria:

* Patients who have previously received any anti-CD19 / anti-CD3 treatment, or any other anti-CD19 treatment;
* Patients previously treated with any gene therapy product, including car-t treatment;
* Patients with detectable cerebrospinal fluid malignant cells or brain metastasis, or patients with a history of central nervous system (CNS) lymphoma or primary CNS lymphoma;
* Patients with testicular invasion, including patients with orchiectomy;
* Patients with current or history of central nervous system diseases, such as epilepsy, cerebrovascular ischemia / hemorrhage, dementia, cerebellar diseases or any autoimmune diseases involving the central nervous system;
* Patients who had previously received allogeneic hematopoietic stem cell transplantation (HSCT);
* Patients who are suitable and willing to receive autologous hematopoietic stem cell transplantation (ASCT);
* The feasibility evaluation screening stage showed that the lymphocyte transfection efficiency of patients was less than 5%, or patients whose T cell culture could not be expanded (< 5 times).
* Patients who received chemotherapy other than lymphocyte clearance chemotherapy within 2 weeks before xkdct023 infusion;
* Patients who had received other study drugs within 30 days before screening;
* Patients who received radiotherapy within 2 weeks before infusion;
* Active hepatitis B (defined as hepatitis B virus DNA detection value > 1000 copies/ml) or hepatitis C virus (HCV RNA positive) patients.
* HIV positive or Treponema pallidum positive patients;
* Patients with acute life-threatening bacterial, viral or fungal infections that have not been controlled (e.g. positive blood culture ≤ 72 hours before infusion);
* Patients with unstable angina pectoris and / or myocardial infarction within 6 months before screening;
* Patients with previous or concurrent malignancies, with the following exceptions: well treated basal cell or squamous cell carcinoma (sufficient wound healing is required before enrollment in the study); Cervical cancer or breast cancer in situ cancer, after curable treatment, had no recurrence at least 3 years before the study. The primary malignant tumor has been completely removed and completely relieved for ≥ 5 years.
* Pregnant or lactating female patients (women of childbearing age are verified as positive results by serum or urine pregnancy test during the screening period);
* There are arrhythmia patients without medical management control;
* Patients who received oral anticoagulant therapy within 1 week before car-t cell infusion;
* Patients who had previously received any adoptive T cell therapy;
* active neuroautoimmune or inflammatory disorders (e.g. Guillian Barre syndrome, amyotrophic lateral sclerosis).

Ages: 18 Days to 75 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Adverse event | The follow-up visit within 2 months is allowed to have a time window of ± 2 days, and the follow-up visit from the 3rd to 12th months is allowed to have a time window of ± 5 days.
  Type, incidence and severity of adverse events
Maximum tolerated dose | The follow-up visit within 2 months is allowed to have a time window of ± 2 days, and the follow-up visit from the 3rd to 12th months is allowed to have a time window of ± 5 days.
  The maximum dose that does not cause death of the subject
Recommended dose for phase II | The follow-up visit within 2 months is allowed to have a time window of ± 2 days, and the follow-up visit from the 3rd to 12th months is allowed to have a time window of ± 5 days.
  Determine the recommended dose for phase II clinical trials

SECONDARY OUTCOMES:
Peak time,Tmax | The follow-up visit within 2 months is allowed to have a time window of ± 2 days, and the follow-up visit from the 3rd to 12th months is allowed to have a time window of ± 5 days.
  Venous blood samples were collected once during the infusion period D1, D2, D4, D6, D8, D10, D12, D14, D16, D18, D21, D24, d27, d30 and follow-up period. The proportion and count of car-t cells in peripheral blood and bone marrow were detected by flow cytometry and RT-PCR, and the PK parameters, PK characteristics and distribution of car-t cells in bone marrow were evaluated. The probe method of fluorescence quantitative PCR was used to monitor the copy number of CAR.
Maximum concentration, Cmax | The follow-up visit within 2 months is allowed to have a time window of ± 2 days, and the follow-up visit from the 3rd to 12th months is allowed to have a time window of ± 5 days.
  Venous blood samples were collected once during the infusion period D1, D2, D4, D6, D8, D10, D12, D14, D16, D18, D21, D24, d27, d30 and follow-up period. The proportion and count of car-t cells in peripheral blood and bone marrow were detected by flow cytometry and RT-PCR, and the PK parameters, PK characteristics and distribution of car-t cells in bone marrow were evaluated. The probe method of fluorescence quantitative PCR was used to monitor the copy number of CAR.
Area Under Curve, AUC1-30d | The follow-up visit within 2 months is allowed to have a time window of ± 2 days, and the follow-up visit from the 3rd to 12th months is allowed to have a time window of ± 5 days.
  Venous blood samples were collected once during the infusion period D1, D2, D4, D6, D8, D10, D12, D14, D16, D18, D21, D24, d27, d30 and follow-up period. The proportion and count of car-t cells in peripheral blood and bone marrow were detected by flow cytometry and RT-PCR, and the PK parameters, PK characteristics and distribution of car-t cells in bone marrow were evaluated. The probe method of fluorescence quantitative PCR was used to monitor the copy number of CAR.
Pharmacodynamics | The follow-up visit within 2 months is allowed to have a time window of ± 2 days, and the follow-up visit from the 3rd to 12th months is allowed to have a time window of ± 5 days.
  The peak value of cytokines within 1 month after car-t cell infusion and the time to return to the baseline state or normal range.
Total remission rate | The follow-up visit within 2 months is allowed to have a time window of ± 2 days, and the follow-up visit from the 3rd to 12th months is allowed to have a time window of ± 5 days.
  The total remission rate of each dose group and all patients evaluated at 1 month, 3 months, 6 months, 9 months and 12 months after car-t treatment.M3 was scanned with systemic CT ± head, neck, chest, abdomen and pelvis enhanced CT. For M6, M9 and M12, enhanced CT or MRI of head, neck, chest and abdominal basin was used.
Complete remission rate | The follow-up visit within 2 months is allowed to have a time window of ± 2 days, and the follow-up visit from the 3rd to 12th months is allowed to have a time window of ± 5 days.
  The complete remission rate of each dose group and all patients evaluated at 1 month, 3 months, 6 months, 9 months and 12 months after car-t treatment.M3 was scanned with systemic CT ± head, neck, chest, abdomen and pelvis enhanced CT. For M6, M9 and M12, enhanced CT or MRI of head, neck, chest and abdominal basin was used.
Partial remission rate | The follow-up visit within 2 months is allowed to have a time window of ± 2 days, and the follow-up visit from the 3rd to 12th months is allowed to have a time window of ± 5 days.
  The partial remission rate of each dose group and all patients evaluated at 1 month, 3 months, 6 months, 9 months and 12 months after car-t treatment.M3 was scanned with systemic CT ± head, neck, chest, abdomen and pelvis enhanced CT. For M6, M9 and M12, enhanced CT or MRI of head, neck, chest and abdominal basin was used.
Distribution of car-t cells in bone marrow | The follow-up visit within 2 months is allowed to have a time window of ± 2 days, and the follow-up visit from the 3rd to 12th months is allowed to have a time window of ± 5 days.
  The proportion and count of car-t cells in peripheral blood and bone marrow were detected by flow cytometry and RT-PCR to evaluate the distribution of car-t cells in bone marrow. The probe method of fluorescence quantitative PCR was used to monitor the copy number of CAR.
Survival of car-t cells | The follow-up visit within 2 months is allowed to have a time window of ± 2 days, and the follow-up visit from the 3rd to 12th months is allowed to have a time window of ± 5 days.
  Survival of car-t cells in adult patients with recurrent or refractory DLBCL.